CLINICAL TRIAL: NCT04614662
Title: Symptom Screening Linked to Care Pathways for Children With Cancer: a Cluster Randomized Trial
Brief Title: Symptom Screening Linked to Care Pathways
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lillian Sung, Pediatric Oncologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1000068699; 1R01CA251112-01 (NIH); PJT-169165 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2020-10-21; First posted 2020-11-04 (Actual); Results first posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Pediatric Cancer; Quality of Life
Keywords: Pediatric Oncology; Cluster Randomized Clinical Trial; Symptom Screening; Quality of Life
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants enrolled at intervention sites will be prompted to complete symptom screening three times weekly via SPARK with corresponding feedback and links to symptom management care pathways sent to their healthcare providers.
  Symptom screening using SPARK can be performed at any time and as often as desired, but screening will be prompted three times weekly for eight weeks.
  Each day the participant completes symptom screening and has at least one severely bothersome symptom, the primary healthcare team will receive an email summarizing the symptom report and highlighting symptoms that are "a lot" or "extremely" bothersome.
  Upon study activation, we will work with each of the 10 intervention sites to develop site-specific, adapted care pathways that consider relevant work flows, institutional culture and available resources.
  Interventions: Behavioral: SPARK Symptom Screening Linked to Feedback to Providers
- Control (No Intervention): At control sites, usual care will be provided, which may or may not include symptom screening, access to CPGs or care pathways. Participants will complete SSPedi to obtain the primary outcome at weeks 0, 4 and 8 but the scores will not be revealed to providers and will not be linked to care pathways.

INTERVENTIONS:
Behavioral: SPARK Symptom Screening Linked to Feedback to Providers — Symptom screening three times weekly via SPARK, feedback of symptoms to healthcare providers and development of care pathways for symptom management.
  Arms: Intervention

SUMMARY:
Most children with cancer survive because they are given intensive treatments, but unfortunately, these treatments are associated with distressing symptoms. To address this problem, we developed the Symptom Screening in Pediatrics Tool (SSPedi) so that children receiving cancer treatments can communicate their bothersome symptoms, and Supportive care Prioritization, Assessment and Recommendations for Kids (SPARK), a web-based application that links identified symptoms to supportive care guidelines for symptom management. To establish that these tools improve the lives of children newly diagnosed with cancer, we will conduct a trial that randomizes 20 pediatric cancer institutions and measures the impact of three times weekly symptom screening, symptom feedback to healthcare providers and the development of care pathways for symptom management to improve total symptom burden, fatigue and quality of life.

DETAILED DESCRIPTION:
Aims 1 and 2: Among children with newly diagnosed cancer, to determine if symptom screening and feedback to healthcare providers at least three times weekly and locally-adapted symptom management care pathways, when compared to usual care:

Aim 1. Improves overall self-reported symptom scores (total SSPedi score), fatigue (PROMIS-Fatigue) and cancer-specific QoL (PedsQL 3.0 Acute Cancer Module) over 8 weeks Hypothesis: Symptom screening and care pathways will improve symptoms, fatigue and QoL

Aim 2. Improves symptom documentation, increases provision of interventions for symptoms, and reduces emergency department visits and unplanned clinic visits and hospitalizations over 8 weeks Hypotheses: Symptom screening and care pathways will increase symptom documentation and provision of interventions for symptoms, and will reduce healthcare utilization.

Aim 3: As an exploratory aim, we will evaluate key elements of the intervention related to the external validity and generalizability of the intervention effects using the RE-AIM framework.

Overall Strategy This is a cluster randomized trial including 20 pediatric oncology sites. The coordinating center is The Hospital for Sick Children in Toronto, Canada. Sites will be randomized to either systematic symptom screening via SPARK with provision of symptom reports to healthcare providers containing links to care pathways for symptom management (intervention) or usual care (control).

Research Methods Eligibility: We will include children with cancer who: (1) are 8-18 years of age at enrollment (SSPedi is validated in this age range); (2) are English or Spanish-speaking (all PROs are validated in these languages in this age range); (3) have any newly diagnosed cancer; (4) have a plan for any chemotherapy, radiotherapy or surgery; and (5) enroll within 28 days after treatment initiation. Exclusion criteria will be cognitive disability (attending lower than second grade or equivalent) or visual impairment (cannot see SPARK even with corrective lens).

Procedures: In this cluster randomized trial, we will randomize sites to either intervention or control groups. At both intervention and control sites, we will enroll participants within 28 days after treatment initiation. Eligible participants will be identified by site personnel and the study will be explained to them by trained research team members. Participant capacity to consent will be assessed by the clinical or research team according to institutional standards. After the study has been explained and sufficient time has been provided to ensure all questions have been answered, informed consent and assent will be obtained from participants and guardians as appropriate. For those who decline to contribute PROs, they will be given the option to only participate in a retrospective chart review to evaluate symptom documentation, intervention provision and healthcare utilization. Careful tracking of all newly diagnosed patients by site research personnel will occur to determine how many patients are approached and consented, and where possible, reasons for declining participation.

For all enrolled participants who will be contributing PROs (excluding those only involved in the retrospective chart review), a personal SPARK account will be created to allow SSPedi to be completed and symptom results to be recorded. At the 10 intervention sites, site-specific symptom management care pathways will be adapted from template care pathways for each of the 15 symptoms included in SSPedi. Enrolled participants will be prompted by text or email to complete symptom screening three times weekly via SPARK with corresponding feedback sent to their healthcare providers. Symptom reports will contain links to care pathways for symptom management. Active intervention will last for eight weeks starting from the date of enrollment. At the 10 control sites, participants will complete SSPedi to obtain the primary outcome at weeks 0, 4 and 8 but the scores will not be revealed to providers and will not be linked to care pathways. Usual care will be provided to participants at control sites and thus, there will be no study-requested routine, systematic symptom screening, symptom feedback to providers, or linkage to care pathways. If sites already routinely perform systematic symptom screening or use care pathways for symptom management, these may be continued but their use will be recorded.

At both intervention and control sites, demographic information including age, sex, race, ethnicity, diagnosis, cancer stage, family socioeconomic information and treatment plan will be collected at enrollment. The following PROs will be obtained by trained research staff at baseline, week 4 and week 8 for all participants: SSPedi, PROMIS Fatigue and the PedsQL 3.0 Acute Cancer Module (Aim 1). We will contact participants ahead of time to coordinate the week 4 and 8 PROs so that they can be completed in person during hospitalizations or clinic visits. If unable to arrange completion of these PROs in person, we will use their contact information to complete the questionnaires by email, text or over the phone. Data from health records (Aim 2) will be abstracted for all enrolled participants. Relapse and cancer treatment received information will be collected at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* 8-18 years of age at enrollment
* English or Spanish-speaking
* Any newly diagnosed cancer
* Have a plan for any chemotherapy, radiotherapy or surgery
* Enroll within 28 days after treatment initiation

Exclusion Criteria:

* Cognitive disability (attending minimum second grade or equivalent)
* Visual impairment (cannot see SPARK even with corrective lens)

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 445 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Sung, MD, PhD, Principal Investigator — The Hospital for Sick Children; Laura Lee Dupuis, RPh, PhD, Principal Investigator — The Hospital for Sick Children; Allison Grimes, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (21):
- United States (20):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - The Leland Stanford Junior University, Redwood City, California
  - University of Colorado Denver, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Nemours Children's Hospital, Delaware, Wilmington, Delaware
  - Nemours Children's Health, Jacksonville, Jacksonville, Florida
  - Nemours Children's Hospital, Florida, Orlando, Florida
  - Kapi'olani Medical Center for Women & Children, Honolulu, Hawaii
  - Unity Point Health - Blank Children's Hospital, Des Moines, Iowa
  - The University of Iowa, Iowa City, Iowa
  - Children's Hospital, New Orleans, Louisiana
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - The Trustees of Columbia University in the City of New York, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - The University of Texas M. D. Anderson Cancer Center, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The full data set including the patient-reported outcome data will be available publically following trial completion after ensuring that no patient can be identified and no disclosure of personal health information. The data will become available no later than one year after the primary publication and will be available for at least five years.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Five years
Access Criteria: Upon request to, and approval by the study team

REFERENCES:
- [Background] Dupuis LL, Johnston DL, Baggott C, Hyslop S, Tomlinson D, Gibson P, Orsey A, Dix D, Price V, Vanan M, Portwine C, Kuczynski S, Spiegler B, Tomlinson GA, Sung L. Validation of the Symptom Screening in Pediatrics Tool in Children Receiving Cancer Treatments. J Natl Cancer Inst. 2018 Jun 1;110(6):661-668. doi: 10.1093/jnci/djx250. PMID 29272441
- [Background] Hinds PS, Nuss SL, Ruccione KS, Withycombe JS, Jacobs S, DeLuca H, Faulkner C, Liu Y, Cheng YI, Gross HE, Wang J, DeWalt DA. PROMIS pediatric measures in pediatric oncology: valid and clinically feasible indicators of patient-reported outcomes. Pediatr Blood Cancer. 2013 Mar;60(3):402-8. doi: 10.1002/pbc.24233. Epub 2012 Jul 24. PMID 22829446
- [Background] Varni JW, Burwinkle TM, Katz ER, Meeske K, Dickinson P. The PedsQL in pediatric cancer: reliability and validity of the Pediatric Quality of Life Inventory Generic Core Scales, Multidimensional Fatigue Scale, and Cancer Module. Cancer. 2002 Apr 1;94(7):2090-106. doi: 10.1002/cncr.10428. PMID 11932914
- [Derived] Dupuis LL, Vettese E, Aftandilian C, Agarwal V, Baggott C, Bradfield SM, Crellin-Parsons N, Freyer DR, Kelly KM, King AA, Kyono W, Nagasubramanian R, Orgel E, Roth ME, Sherani F, Yu L, Grimes AC, Beauchemin MP, Klesges LM, Tomlinson GA, Sung L. Factors Associated With Self-Report Symptom Screening Adherence in Pediatric Cancer Patients. Cancer Med. 2025 Jul;14(14):e71053. doi: 10.1002/cam4.71053. PMID 40686265
- [Derived] Dupuis LL, Vettese E, Grimes AC, Beauchemin MP, Klesges LM, Baggott C, Demedis J, Aftandilian C, Freyer DR, Crellin-Parsons N, Orgel E, Dickens D, Kelly KM, Kyono W, Walsh A, Sherani F, Cannone D, Orsey AD, King AA, Yu L, Woods-Swafford W, Bradfield SM, Roth ME, Esbenshade AJ, Caywood EH, Agarwal V, Nagasubramanian R, Tomlinson GA, Sung L. Symptom Screening Linked to Care Pathways for Pediatric Patients With Cancer: A Randomized Clinical Trial. JAMA. 2024 Dec 17;332(23):1981-1991. doi: 10.1001/jama.2024.19585. PMID 39535768
- [Derived] Vettese E, Sherani F, King AA, Yu L, Aftandilian C, Baggott C, Agarwal V, Nagasubramanian R, Kelly KM, Freyer DR, Orgel E, Bradfield SM, Kyono W, Roth M, Klesges LM, Beauchemin M, Grimes A, Tomlinson G, Dupuis LL, Sung L. Symptom management care pathway adaptation process and specific adaptation decisions. BMC Cancer. 2023 Apr 17;23(1):350. doi: 10.1186/s12885-023-10835-0. PMID 37069510
- [Derived] Dupuis LL, Grimes A, Vettese E, Klesges LM, Sung L. Readiness to Implement Symptom Management Care Pathways in Pediatric Cancer. Res Sq [Preprint]. 2020 Dec 30:rs.3.rs-136225. doi: 10.21203/rs.3.rs-136225/v1. PMID 33398260

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Pediatric Healthcare Sites
Groups:
- Intervention: Participants enrolled at intervention sites will be prompted to complete symptom screening three times weekly via SPARK with corresponding feedback and links to symptom management care pathways sent to their healthcare providers.
  Symptom screening using SPARK can be performed at any time and as often as desired, but screening will be prompted three times weekly for eight weeks.
  Each day the participant completes symptom screening and has at least one severely bothersome symptom, the primary healthcare team will receive an email summarizing the symptom report and highlighting symptoms that are "a lot" or "extremely" bothersome.
  Upon study activation, we will work with each of the 10 intervention sites to develop site-specific, adapted care pathways that consider relevant work flows, institutional culture and available resources.
  SPARK Symptom Screening Linked to Feedback to Providers: Symptom screening three times weekly via SPARK, feedback of symptoms to healthcare providers and development of care pathways for symptom management.
Period: Overall Study
Arm/Group | Control | Intervention
Started | 224; 10 Pediatric Healthcare Sites | 221; 10 Pediatric Healthcare Sites
Completed | 224; 10 Pediatric Healthcare Sites | 220; 10 Pediatric Healthcare Sites
Not Completed | 0; 0 Pediatric Healthcare Sites | 1; 0 Pediatric Healthcare Sites
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 221 | 224 | 445
Age, Customized [Number; unit: Participants] — Minimum = 8, Maximum = 18
  Participants
    8-10 | 33 | 37 | 70
    11-14 | 77 | 85 | 162
    15-18 | 111 | 102 | 213
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 95 | 183
  Male | 133 | 129 | 262
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 85 | 63 | 148
  Not Hispanic or Latino | 123 | 139 | 262
  Unknown or Not Reported | 13 | 22 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 4 | 6
  Asian | 13 | 7 | 20
  Native Hawaiian or Other Pacific Islander | 14 | 1 | 15
  Black or African American | 13 | 14 | 27
  White | 113 | 145 | 258
  More than one race | 22 | 12 | 34
  Unknown or Not Reported | 44 | 41 | 85
Baseline total SSPedi Score [Mean (Standard Deviation); unit: sum of the 15 SSPedi items' scores] — SSPedi scale per item: 0 (Not at all bothered) to 4 (Extremely bothered)
  Minimum SSPedi score: 0, Maximum SSPedi score: 60, where a higher score indicates a worse outcome.
  sum of the 15 SSPedi items' scores | 11.8 (8.2) | 13.5 (8.2) | 12.7 (8.2)

OUTCOME MEASURES:

1. Primary Outcome: Symptom Screening in Pediatrics Tool (SSPedi) Total Score
Description: SSPedi measures the degree to which 15 symptoms bothered the participant yesterday or today. Each symptom is scored on a 5-point Likert scale ranging from 0 (not at all bothered) to 4 (extremely bothered). The total score ranges from 0 to 60 where higher numbers indicate more bothersome symptoms. The total SSPedi score is reliable, valid and responsive to change in children with cancer 8-18 years of age.(1)
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 198 | 213
Score on a scale | 7.9 (7.2) | 11.4 (8.7)

2. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Bank v2.0 - Fatigue
Description: Fatigue will be measured using PROMIS. PROMIS uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation of that population. The minimum raw score for this measure is 10 and the maximum raw score is 50. The recall period is the last 7 days and a higher score equals more fatigue. It is reliable and valid in children 8-18 years of age with cancer. This was administered using CAT (Computer Adaptive Test) scoring through REDCap. With a CAT, participant responses guide the system's choice of subsequent items from the full item bank. As additional items are administered, the potential for error is reduced and confidence in the respondent's score increases. T score conversion table 'PROMIS - Fatigue 10a Pediatric' was used.
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Control | Intervention
Number analyzed (Participants) | 224 | 221
T score | 54.6 (12.1) | 53.9 (12.1)

3. Secondary Outcome: PedsQL 3.0 Acute Cancer Module
Description: This is a cancer-specific measure of quality of life. It assesses pain and hurt, nausea, procedural anxiety, treatment anxiety, worry, cognitive problems, perceived physical appearance and communication. The self-report 7-day recall version will be used. The minimum value on the scale is 0 and maximum value is 100. PedsQL uses reverse scoring thus a higher score indicates a better outcome. Each question uses a Likert scale ranging from 0 to 4 for raw scores, and 0 to 100 for scaled scores. The breakdown of items per domain is as follows: Pain and Hurt: 2 items, Nausea: 5 items, Procedural Anxiety, Treatment Anxiety, Worry, Perceived Physical Appearance and Communication: 3 items each, Cognitive Problems: 4 items. Scaled items from each subscale are averaged to create a final score, where a higher score indicates a better outcome.
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 224 | 221
units on a scale
  PedsQL 3.0 domain score: Pain and hurt | 68.8 (24.8) | 69.8 (26.6)
  PedsQL 3.0 domain score: Nausea | 69.2 (20.7) | 73.9 (23.4)
  PedsQL 3.0 domain score: Procedural anxiety | 62.8 (29.1) | 66.4 (30.3)
  PedsQL 3.0 domain score: Treatment anxiety | 76.0 (23.4) | 77.7 (26.3)
  PedsQL 3.0 domain score: Worry | 62.8 (22.8) | 64.7 (26.6)
  PedsQL 3.0 domain score: Cognitive problems | 69.1 (20.6) | 70.3 (21.2)
  PedsQL 3.0 domain score: Perceived physical appearance | 73.2 (26.4) | 74.7 (25.0)
  PedsQL 3.0 domain score: Communication | 73.2 (21.7) | 77.8 (21.3)

4. Secondary Outcome: Documentation of Symptoms
Description: This outcome will be obtained with a one day window before and after the week 8 patient-reported outcome assessment. The number below represents participants with instances of symptom documentation. Documentation means there was some notation in the medical record of that symptom.
Time Frame: Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 224 | 221
Participants
  Feeling dissapointed or sad | 28 | 16
  Feeling scared or worried | 40 | 26
  Feeling cranky or angry | 9 | 7
  Problems with thinking or remembering things | 2 | 3
  Changes in how your body or face look | 8 | 5
  Feeling tired | 61 | 43
  Mouth sores | 8 | 8
  Headache | 19 | 15
  Hurt or pain | 46 | 57
  Tingly or numb hands or feet | 15 | 15
  Throwing up or feeling like you may throwup | 62 | 58
  Feeling more or less hungry than you usually do | 37 | 22
  Changes in taste | 2 | 7
  Constipation | 15 | 20
  Diarrhea | 3 | 6

5. Secondary Outcome: Provision of Interventions for Symptoms (Independent of Symptom Documentation)
Description: The number of interventions for each symptom at each reporting period will be recorded and categorized as any intervention provided vs. no intervention provided. Interventions included in the local care pathway will be noted. This outcome will be obtained with a one day window after the week 8 patient-reported outcome assessment. Any intervention regardless of attribution was abstracted from a list of potential, previously-defined interventions for specific symptoms. For example a child life specialist visit was considered an intervention for sadness, anxiety and anger, regardless of visit reason. Interventions for symptoms are recorded regardless of whether a symptom was documented in the chart, for example, acetaminophen was considered an intervention for pain, even if there was no documentation of pain reported. The numbers listed below represent the count of participants with any interventions provided, regardless of documentation for the symptom being recorded.
Time Frame: Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 221 | 224
Participants
  Feeling dissapointed or sad | 52 | 82
  Feeling scared or worried | 54 | 96
  Feeling cranky or angry | 48 | 67
  Problems with thinking or remembering things | 5 | 5
  Changes in how your body or face look | 0 | 1
  Feeling tired | 12 | 15
  Mouth sores | 28 | 23
  Headache | 35 | 42
  Hurt or pain | 68 | 70
  Tingly or numb hands or feet | 17 | 25
  Throwing up or feeling like you may throw up | 119 | 134
  Feeling more or less hungry than you usually do | 18 | 20
  Changes in taste | 2 | 0
  Constipation | 59 | 57
  Diarrhea | 0 | 1

6. Secondary Outcome: Number of Emergency Department Visits and Unplanned Clinic Visits and Hospitalizations
Description: Number of visits to the emergency room and unplanned clinic visits and hospitalizations will be summed over the 8 week on-study period.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Unplanned Health Care Encounters
Arm/Group | Intervention | Control
Number analyzed (Participants) | 221 | 224
Unplanned Health Care Encounters | 1.82 (2.34) | 1.12 (1.62)

ADVERSE EVENTS:
Time Frame: 8 weeks; Adverse events were monitored for the duration of the study with enrolled participants (August 2, 2021 - October 18, 2023)
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/221 | 0/224
Serious Adverse Events (participants affected / at risk) | 0/221 | 0/224
Other Adverse Events (participants affected / at risk) | 0/221 | 0/224

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-11-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT04614662/Prot_002.pdf
  • Statistical Analysis Plan (2023-11-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT04614662/SAP_001.pdf